CLINICAL TRIAL: NCT07210125
Title: Implementation and Delivery of Lenacapavir for PrEP in a Community Pharmacy Setting
Brief Title: Implementation and Deliver of Lenacapavir for PrEP in a Community Pharmacy Setting
Acronym: L4PinPharm
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kelley-Ross & Associates, Inc. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IN-US-974-7746
Record Dates: First submitted 2025-09-15; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: HIV PrEP; Lenacapavir; Pharmacist-managed PrEP,; L4P; Pre-exposure prophylaxis; community pharmacy PrEP
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Aim 1 is a prospective observational study enrolling 75 subjects into the cohort to report on the feasibility and acceptability of a pharmacist-managed L4P in a community pharmacy setting. Aim 2 is a retrospective matched cohort study to assess the differences in retention and STI positivity rates between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AIM 1: lenacapavir for PrEP managed by pharmacists (Experimental): prospective observational study enrolling 75 subjects into the cohort to report on the feasibility and acceptability of a pharmacist-managed L4P in a community pharmacy setting. This will be done as a longitudinal, observational, mixed methods study to report on experiences of operating this service for 1 year.
  Interventions: Drug: Lenacapavir long-acting
- AIM 2: retrospective cohort study to assess the impact on PrEP visits every 3 months vs. every 6 mon (Experimental): The 75 subjects who provided informed consent will be retrospectively case control matched to a cohort of people for age, gender identity, insurance status, postal code, predictors of STI risk, number of partners, genders of partners, condomless sex, receptive anal sex. Adjustments will be made to matching ratio if all matches are not found.
  Interventions: Drug: Lenacapavir long-acting; Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Lenacapavir long-acting — Until recently, only oral formulations of PrEP were available. With the availability of long-acting PrEP injectables, new strategies will need to be developed to deliver this new treatment option. The availability of L4P offers an opportunity to expand PrEP access outside traditional healthcare settings. However, data on the feasibility and acceptability of L4P in community pharmacies is lacking. Community pharmacies are ideal for L4P due to their accessibility and the ability to utilize both pharmacy and medical billing for reimbursement of medication and clinical services, unlike traditional healthcare settings. Pharmacists are one of the most highly accessible healthcare professionals in the community. There are over 60,000 community pharmacies across the U.S. The study will evaluate implementation outcomes (feasibility, acceptability), real-world effectiveness, and whether L4P can be used for same day starts or treatment switches.
Other: Standard of Care (SOC) — In aim 2, subjects enrolled in the L4P cohort will have the option of conducting STI testing every 6 months versus every 3 months. A retrospective matched cohort study will be conducted to assess the differences in retention and STI positivity rates between groups. All participants will be able to get tested in between monitoring visits.
  Arms: AIM 2: retrospective cohort study to assess the impact on PrEP visits every 3 months vs. every 6 mon

SUMMARY:
This is an open-label, single center study to evaluate implementation of a pharmacist-managed delivery of L4P in a community pharmacy setting and the impact of twice-yearly vs. quarterly PrEP visits on STI rates.

DETAILED DESCRIPTION:
This is a prospective observational study enrolling 75 subjects into the cohort to report on the feasibility and acceptability of a pharmacist-managed L4P in a community pharmacy setting. The study will be conducted as a longitudinal, observational, mixed methods evaluation of the operation of this service for 1 year using existing pharmacy clinic models and infrastructure. The investigators will also conduct a retrospective cohort study to assess the impact on PrEP visits every 3 months versus every 6 months. All subjects must meet all eligibility criteria to participate in the study. Subjects will have the opportunity to start or switch to commercially available L4P. PrEP initiation will be defined as subjects starting PrEP who have not taken PrEP for the previous 3 months. All FDA-approved PrEP products indicated for each individual will be offered, and each patient will have the opportunity to participate in the study. Patients interested in initiating will be offered the opportunity to enroll and provide informed consent. Initiation of L4P will be based on medical, laboratory, and coverage qualifications.

Patients on L4P will be managed by a pharmacist provider utilizing a CDTA based on the DHHS Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents with HIV and the FDA-approved label for lenacapavir. L4P will be administered on Day 1, Day 2 (oral loading dose only), and every six months thereafter. Subjects will be followed for 12 months, and electronic health record data will be collected retrospectively throughout the study duration. Subjects will be given a survey 4 to 6 weeks after initiation and at study end. Subjects will have the option to discontinue participation at any time for any reason, and standards of care for discontinuation will be followed. Participants who do not meet criteria for management under the CDTA (positive HIV screening, pregnancy, or other complicated health conditions) will be referred to an existing primary care provider or the clinic medical director for further management. Referrals for substance use treatment, mental health, and primary care services will also be provided. At the end of the study, each patient will complete a survey and be offered the option to continue commercially available L4P.

L4P will be administered by the pharmacist provider. A pharmacist training program will be created by the study team and completed by all pharmacists providing L4P services. Pharmacies are health care settings, and all safety measures will be followed for the administration of L4P. These measures include informed consent and counseling on risks versus benefits, post-injection observation, policies and procedures in place for emergency services and allergic reactions. Access to epinephrine and diphenhydramine will be onsite. All pharmacist providers will have CPR and blood-borne pathogen training. Pharmacists who enroll in the study and provide informed consent will be given a survey at study start and end. The pharmacist surveys will be validated psychometric assessments measuring implementation outcomes often considered "leading indicators" of implementation success: Acceptability of Intervention (AIM), Intervention Appropriateness Measure (IAM), and Feasibility Intervention Measure (FIM).

A pharmacy technician will assist with administrative tasks such as scheduling, billing, prior authorizations, benefit verification, and patient assistance programs. Specific attention will be given to overcoming billing barriers. Commercial drug product will be utilized in this study. To create a sustainable program after funding ceases, real-world reimbursement programs, such as insurance and patient assistance programs, will be used to reimburse pharmacist time for performing these clinical services and for the reimbursement of commercial drug product. Uninsured patients will have the opportunity to participate. The pharmacy technician will assist patients in enrolling in state and commercial drug assistance programs to cover service and medication costs.

The study intervention is divided into two aims. For Aim 1, the investigators will conduct a prospective observational study enrolling 75 subjects into the cohort to report on the feasibility and acceptability of a pharmacist-managed L4P in a community pharmacy setting. This will be conducted as a longitudinal, observational, mixed methods evaluation of operating this service for 1 year. The primary objective is feasibility as measured by retention. Additional feasibility outcomes include adherence, persistence, and seroconversion collected through EHR review. Secondary outcomes include acceptability (as determined by subject and provider surveys), STI rates, HIV seroconversions, reasons for discontinuation, and pharmacist and patient perspectives on barriers and facilitators. In Aim 2, subjects enrolled in the L4P cohort will have the option of conducting STI testing every 6 months versus every 3 months. A retrospective matched cohort study will be conducted to assess differences in retention and STI positivity rates between groups. All participants will be able to undergo testing in between monitoring visits. The primary outcome measure will be adherence to PrEP medication as measured by the proportion of participants who successfully attend their PrEP monitoring visits over 12 months. Secondary outcomes include visit frequency and STI positivity rate. Visit frequency will be measured as the overall number of PrEP visits and in-between STI visits per person-year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of screening
* weight greater than or equal to 35kg
* HIV-negative status
* Willing to provide informed consent and undergo all required study procedures

Exclusion Criteria:

* Unknown or positive HIV status
* Coadministration of drugs that significantly decreases lenacapavir concentrations according to the FDA package insert
* Any participant that do not meet criteria for management under the CDTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention Rate | 1 year
  Calculated by dividing the number of participants present in the study at 1 year by the number of individuals enrolled
Adherence Rate | 1 year
  Collected as the proportion of injections that are successfully administered during each target injection window period over 1 year
Persistence | 1 year
  Measured as the length of time a person remains on L4P for over 1 year

SECONDARY OUTCOMES:
Patient acceptability of a pharmacist managed L4P service. | 1 year
  Patient Acceptability will be measured by the HIV-PrevTSQs questionnaire at baseline (for those already on an FDA approved PrEP regimen within 3 months from enrollment), 4-6 weeks and 1 year and HIV-PrevTSQc at 1 year. It is a 6 point Likert scale questionnaire which higher scores indicating higher acceptability.
Pharmacist Acceptability of a pharmacist managed L4P service | 1 year
  Assessed using the FIM, AIM, and IAM surveys at baseline and 1 year. These surveys are a 5 point Likert scale with a range of scores from 4-20. The higher the score, the more favorable the perceptions.
Visit Frequency between people receiving PrEP visits every 3 months versus every 6 months. | 1 year
  Visit frequency will be measured as the overall number of PrEP visits and in-between STI visits per person year.
STI Positivity Rates in 6-month versus 3-month PrEP monitoring visits. | 1 year
  Measured as the number of chlamydia, gonorrhea, or syphilis diagnosed per 100 visits.

OTHER OUTCOMES:
L4P initiations | 1 year
  Number of L4P starts by end of 1 year
Time to first injection | 1 year
  Time it takes to get from enrollment to first injection
HIV seroconversions | 1 year
  Rate of HIV infections at the end of 1 year
STI Rates | 1 year
  Rate of STI infections (chlamydia, gonorrhea, or syphilis) at the end of 1 year
Reasons for discontinuation | 1 year
  collect verbally or written reasons for early discontinuation
Adverse Reactions | 1 year
  rates of adverse reactions at the end of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kelley-Ross Pharmacy, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data underlying the results will be shared upon reasonable request after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after last patient, last visit for 1 year, for 1 year
Access Criteria: Access will be granted following review of a written proposal and execution of a data use agreement
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Background] Groot Bruinderink ML, Boyd A, Coyer L, Boers S, Blitz L, Brand JM, Gotz HM, Stip M, Woudstra J, Yap K, Vermey K, Matser A, Feddes AR, Jongen VW, Prins M, Hoornenborg E, van Harreveld F, Schim van der Loeff MF, Davidovich U. Online-Mediated HIV Pre-exposure Prophylaxis Care and Reduced Monitoring Frequency for Men Who Have Sex With Men: Protocol for a Randomized Controlled Noninferiority Trial (EZI-PrEP Study). JMIR Res Protoc. 2023 Nov 8;12:e51023. doi: 10.2196/51023. PMID 37938875
- See also: Centers for Disease Control and Prevention. Advancing team based care through collaborative practice agreements: a resource and implementation guide for adding pharmacists to the care team. Atlanta, GA, USA: Centers for Disease Control and Prevention, U. — https://www.cdc.gov/cardiovascular-resources/media/cpa-team-based-care.pdf
- See also: Gilead Sciences, Inc. (n.d.). Yetztugo™ (lenacapavir) tablets for oral use: Prescribing information — https://www.gilead.com/-/media/files/pdfs/medicines/hiv/yeztugo/yeztugo_pi.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT07210125/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT07210125/ICF_001.pdf